CLINICAL TRIAL: NCT03989700
Title: Effect of Thiamin Supplementation on Thiamin Status in Children With Heart Disease Receiving Diuretic Drugs: Randomized Controlled Trial
Brief Title: Effect of Thiamin Supplementation on Thiamin Status in Children With Heart Disease Receiving Diuretic Drugs
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Narumon Densupsoontorn, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si364/2019
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Heart Diseases
Keywords: Diuretic drugs; Thiamin deficiency
MeSH Terms: conditions — Heart Diseases; Beriberi | interventions — Thiamine

STUDY DESIGN:
Intervention Model Description: 1. Enroll children with heart disease receiving diuretic drugs
  2. Evaluate thiamin status by measuring thiamin pyrophosphate effect, cardiac function by echocardiography
  3. Randomize subjects into 3 arms: 2 groups receive different dosages of thiamin supplementation and 1 group receives placebo for 4 weeks
  4. After 4 weeks, thiamin status and echocardiography are evaluated.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): Low dose of thiamin supplementation
  Interventions: Drug: Thiamine Mononitrate
- High dose (Experimental): High dose of thiamin supplementation
  Interventions: Drug: Thiamine Mononitrate
- Placebo (Placebo Comparator): placebo supplementation
  Interventions: Drug: Thiamine Mononitrate

INTERVENTIONS:
Drug: Thiamine Mononitrate — Low dose group: thaimine mononitrate 25 mg/day per oral daily for 4 weeks High dose group: thaimine mononitrate 50 mg/day per oral daily for 4 weeks Placebo group: placebo 25 mg/day per oral daily for 4 weeks
  Other Names: Vitamin B1

SUMMARY:
The purpose of this study is to determine effect of thiamin supplementation on thiamin status by measuring thiamin pyrophosphate effect in children with heart disease receiving diuretic drugs.

DETAILED DESCRIPTION:
Children with heart disease receiving diuretic drugs are susceptible to thiamin deficiency due to increase renal loss. Thiamin deficiency causes abnormal cardiac contraction resulting in heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month old to 15 years old diagnosed as heart disease
* Receiving diuretic drugs at least 1 month

Exclusion Criteria:

* Receiving thiamin-containing vitamins
* Receiving hemodialysis or peritoneal dialysis
* Having problems of intestinal malabsorption, chronic lung disease, red blood cell abnormality such as thalassemia , abnormal hemoglobin typing, G6PD deficiency
* Receiving thiamin-producing probiotics
* Receiving inotropic drugs
* Severe anemia: Hb < 7 g/dL

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in thiamin pyrophosphate effect | 4 weeks
  Compare percentage change in thiamin pyrophosphate effect before and after thiamin supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Narumon Densupsoontorn, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiNicolantonio JJ, Niazi AK, Lavie CJ, O'Keefe JH, Ventura HO. Thiamine supplementation for the treatment of heart failure: a review of the literature. Congest Heart Fail. 2013 Jul-Aug;19(4):214-22. doi: 10.1111/chf.12037. PMID 23910704
- [Background] Katta N, Balla S, Alpert MA. Does Long-Term Furosemide Therapy Cause Thiamine Deficiency in Patients with Heart Failure? A Focused Review. Am J Med. 2016 Jul;129(7):753.e7-753.e11. doi: 10.1016/j.amjmed.2016.01.037. Epub 2016 Feb 18. PMID 26899752
- [Background] Suter PM, Vetter W. Diuretics and vitamin B1: are diuretics a risk factor for thiamin malnutrition? Nutr Rev. 2000 Oct;58(10):319-23. doi: 10.1111/j.1753-4887.2000.tb01827.x. PMID 11127971
- [Background] Brady JA, Rock CL, Horneffer MR. Thiamin status, diuretic medications, and the management of congestive heart failure. J Am Diet Assoc. 1995 May;95(5):541-4. doi: 10.1016/S0002-8223(95)00148-4. PMID 7722187
- [Background] Zenuk C, Healey J, Donnelly J, Vaillancourt R, Almalki Y, Smith S. Thiamine deficiency in congestive heart failure patients receiving long term furosemide therapy. Can J Clin Pharmacol. 2003 Winter;10(4):184-8. PMID 14712323
- [Background] Shamir R, Dagan O, Abramovitch D, Abramovitch T, Vidne BA, Dinari G. Thiamine deficiency in children with congenital heart disease before and after corrective surgery. JPEN J Parenter Enteral Nutr. 2000 May-Jun;24(3):154-8. doi: 10.1177/0148607100024003154. PMID 10850940
- [Background] Schoenenberger AW, Schoenenberger-Berzins R, der Maur CA, Suter PM, Vergopoulos A, Erne P. Thiamine supplementation in symptomatic chronic heart failure: a randomized, double-blind, placebo-controlled, cross-over pilot study. Clin Res Cardiol. 2012 Mar;101(3):159-64. doi: 10.1007/s00392-011-0376-2. Epub 2011 Nov 5. PMID 22057652
- [Background] Shimon I, Almog S, Vered Z, Seligmann H, Shefi M, Peleg E, Rosenthal T, Motro M, Halkin H, Ezra D. Improved left ventricular function after thiamine supplementation in patients with congestive heart failure receiving long-term furosemide therapy. Am J Med. 1995 May;98(5):485-90. doi: 10.1016/s0002-9343(99)80349-0. PMID 7733128
- [Background] Yui Y, Itokawa Y, Kawai C. Furosemide-induced thiamine deficiency. Cardiovasc Res. 1980 Sep;14(9):537-40. doi: 10.1093/cvr/14.9.537. PMID 7214397
- [Background] LeBlanc JG, Chain F, Martin R, Bermudez-Humaran LG, Courau S, Langella P. Beneficial effects on host energy metabolism of short-chain fatty acids and vitamins produced by commensal and probiotic bacteria. Microb Cell Fact. 2017 May 8;16(1):79. doi: 10.1186/s12934-017-0691-z. PMID 28482838
- [Background] Rogovik AL, Vohra S, Goldman RD. Safety considerations and potential interactions of vitamins: should vitamins be considered drugs? Ann Pharmacother. 2010 Feb;44(2):311-24. doi: 10.1345/aph.1M238. Epub 2009 Dec 29. PMID 20040703